CLINICAL TRIAL: NCT03911206
Title: The Duke Healthy Breathing Study Stage 2 (DHBS): A Randomized Controlled Trial Assessing the Safety and Feasibility of Respiratory Muscle Training and Exercise Training in Children and Adolescents With Persistent Asthma
Brief Title: A Trial Assessing the Safety and Feasibility of Respiratory Muscle Training and Exercise Training in Children and Adolescents With Persistent Asthma
Acronym: DHBS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00100666
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 : Inspirtory muscle training (IMT) (Experimental): IMT exercises at home will gradually ramp up.
  Interventions: Behavioral: Inspiratory muscle training (IMT)
- Arm 2: Exercise alone (Experimental): Subjects will be asked to exercise 2x/week for 6 weeks in person at the Duke research facility and again 2x/week at home for 30 minutes.
  Interventions: Behavioral: Exercise alone
- Arm 3: IMT and Exercise (Experimental): a combination of arm 1 and arm 3
  Interventions: Behavioral: IMT and Exercise
- Arm 4: Routine care (No Intervention): no interventions will occur in this group besides testing procedures and offering access to the study team in case asthma-related questions come up.

INTERVENTIONS:
Behavioral: Inspiratory muscle training (IMT) — IMT exercises at home will gradually ramp up
  Arms: Arm 1 : Inspirtory muscle training (IMT)
Behavioral: Exercise alone — Subjects will be asked to exercise 2x/week for 6 weeks in person at the Duke research facility and again 2x/week at home for 30 minutes.
  Arms: Arm 2: Exercise alone
Behavioral: IMT and Exercise — Combining IMT training and exercise
  Arms: Arm 3: IMT and Exercise

SUMMARY:
The purpose of this study is to assess the safety and tolerability of a 6-week Inspiratory Muscle Training and cardiovascular exercise training program in children and adolescents with asthma.

To also determine the efficacy of inspiratory muscle training and exercise in increasing respiratory muscle strength and endurance, and to explore relationships between fitness interventions (inspiratory muscle training and exercise), exercise tolerance, airway closure and dyspnea scores.

ELIGIBILITY:
Inclusion Criteria:

* 10-17 years of age
* Clinician-diagnosed asthma
* Sedentary activity defined as having not participated in a sports team or formal activity (dance classes, gym membership, active hobby requiring physical activity) in the past 12 months or have a
* Body mass index (BMI) ≥85th percentile (adjusted for sex and age)
* Child must have a designated caregiver who expresses a commitment to encourage the participant to attend weekly clinic-based exercise and also complete additional home exercise.

Exclusion Criteria:

* Previous intubation for asthma,
* Forced expiratory volume in 1 second (FEV1) < 50% of predicted at enrollment;
* Any major chronic illness that in the opinion of the PI would interfere with participation in the intervention or completion of the study procedures;
* Inability to complete baseline measurements in a satisfactory manner according to the judgment of the research coordinator or PI
* Currently active in sports, vigorous play or planned exercise more than 1 time per week on average over the past month
* Current Pregnancy as determined by urine pregnancy test.
* Parent/Caregiver unable to consent in English

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participant's with asthma and not participating in any physical activity | 6 weeks
Number of Adverse events reported by participants. | 6 weeks
Number of participants that complete respiratory muscle training (IMT) and exercise. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No